CLINICAL TRIAL: NCT04066712
Title: A Phase 1, Open-Label, Multiple-Dose Study to Evaluate the Pharmacokinetics and Pharmacodynamics of LC350189 in Subjects With Varying Degrees of Renal Impairment
Brief Title: Renal PK Study of LC350189
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-GDCL003
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2019-11

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A: Normal (control) renal function (Experimental)
  Interventions: Drug: LC350189 200 mg
- B: Mild impairment renal function (Experimental)
  Interventions: Drug: LC350189 200 mg
- C: Moderate impairment renal function (Experimental)
  Interventions: Drug: LC350189 200 mg
- D: Severe impairment renal function (Experimental)
  Interventions: Drug: LC350189 200 mg

INTERVENTIONS:
Drug: LC350189 200 mg — Study drug in capsule form, take two capsules of LC350189 100mg, by oral, once daily, from Day 1 through 7

SUMMARY:
This is a Phase 1, open-label, parallel-group, multiple-dose study designed to assess the effect of renal impairment on the PK and PD of LC350189.

ELIGIBILITY:
Inclusion Criteria

* The subject has a BMI of 18 to 40 kg/m2, inclusive, at screening.
* The subject is able to provide written informed consent.

For healthy subjects only : The subject has normal renal function as determined by eGFR and calculated using the MDRD formula, or by 24-hour urine creatinine clearance (CLcr) corrected for body size.

For subjects with renal impairment only

: The subject has mild, moderate, or severe renal impairment as determined by eGFR and calculated using the MDRD formula.

Exclusion Criteria

* The subject has a history or clinical manifestations of a significant neurological, cardiovascular, endocrine, gastrointestinal, pulmonary, hematologic, immunologic, or psychiatric disease that would preclude study participation, as judged by the investigator.
* The subject has nephrotic syndrome, defined as serum albumin <3.0 g/dL and urine protein/creatinine ratio >350 mg/mmol (as an estimate of approximate proteinuria of >3.5 g/day) at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
AUC from time 0 to the last quantifiable concentration | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
AUC from time 0 to 24 hours post dose | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
AUC from time 0 to the end of the dosing interval at steady state | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
Maximum observed plasma concentration | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
Maximum observed plasma concentration at steady state | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
Time to reach maximum observed plasma concentration | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
Time to reach maximum observed plasma concentration at steady state | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments
Amount of drug excreted in urine (Ae) over each collection interval | Before dosing on Days 1 through Day 8
  Pharmacokinetic Assessments

SECONDARY OUTCOMES:
Serum mean concentration over 24 hours | Before dosing on Days 1 through Day 8
  Pharmacodynamic Assessments (uric acid, xanthine, and hypoxanthine)
Maximum observed effect | Before dosing on Days 1 through Day 8
  Pharmacodynamic Assessments (uric acid, xanthine, and hypoxanthine)
Time to reach maximum effect | Before dosing on Days 1 through Day 8
  Pharmacodynamic Assessments (uric acid, xanthine, and hypoxanthine)
Incidence of adverse events | Days 1 through Day 9 (end of study)
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided